CLINICAL TRIAL: NCT03346395
Title: A Problem Solving Based Intervention in Primary Health Care for Facilitating Return-to-work Among People Suffering From Common Mental Disorders - a Cluster-randomized Trial
Brief Title: A Problem Solving Based Intervention for Facilitating Return-to-work Among People Suffering From Common Mental Disorders
Acronym: PROSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Elisabeth Björk Brämberg, PhD, Associate professor, docent, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-07415
Record Dates: First submitted 2017-10-11; First posted 2017-11-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anxiety Disorders; Adjustment Disorders; Common Mental Disorder
Keywords: Adjustment disorders; Anxiety disorders; Depression; Mental disorders; Interventional study; Primary health care; Problem solving; Randomized controlled trial; Return to work; Sick leave
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem solving based intervention (Experimental): The problem solving based intervention contains a problem solving process and cooperation between the person on sick leave, his/her employer and health care professionals. The intervention consists of five steps: 1) Making an inventory of problems and/or opportunities related to return to work; 2) brainstorming about solutions; 3) writing down solutions, identifying the support needed to implement the solutions; 4) a three-party meeting with the person on sick leave, his/her employer and the rehabilitation coordinator; 5) evaluation of the action plan and implementation of solutions, relapse prevention. The intervention takes the form of two to five consultations. The first and fourth steps are key elements.
  Interventions: Behavioral: Problem solving based intervention
- Care as usual (Active Comparator): Medical treatment, or behavioral therapy or in combination. Meeting with a rehabilitation coordinator if that is a part or care as usual within primary health care.
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Problem solving based intervention — Problem solving based intervention
  Arms: Problem solving based intervention
Behavioral: Care as usual — Medical treatment, or behavioral therapy or a coordination of behavioral therapy and medical treatment. Meeting with a rehabilitation coordinator.
  Arms: Care as usual

SUMMARY:
Problem solving based intervention involving the workplace has shown promising effects on return-to-work among persons with common mental disorders. A key element is cooperation between the person on sick leave, the participant's employer and health care professionals. The aim of the present study is to evaluate the effects of a problem solving based intervention in the Swedish primary health care system on an employed population on sick leave due to common mental disorders. Cluster randomized controlled trial. The investigators hypothesize that:

Participants who have undergone the work-related problem solving based intervention will have fewer total days on sick leave than the participants who receive treatment as usual at 18 months.

Participants who receive the work-related problem solving based intervention will have fewer recurrent periods of sick leave than the participants who receive treatment as usual at 18 months.

Participants who receive the work-related problem solving therapy intervention will score better on the secondary outcomes than the participants in the control group.

Population: Employed, aged 18 - 59, on short-term sick leave (min. 2 - max. 12 weeks) due to common mental disorders.

Intervention: Work-related problem solving based intervention in addition to treatment as usual. The intervention will be given by rehabilitation coordinators on max. five occasions and includes: making an inventory of problems and/or opportunities related to return-to-work; identifying the support needed to implement the solutions; a meeting with the person on sick leave, his/her employer and the rehabilitation coordinator to discuss solutions; making an action plan and evaluation.

Control: The control group will receive care as usual (i.e. cognitive behavioral therapy and/or medical treatment, and meeting with a rehabilitation coordinator if this is a part of care as usual at the primary health care centre). A total of 220 persons on sick leave and 30 rehabilitation coordinators will be included.

Primary outcome: total number of days on sick leave at 18 months after baseline. A parallel process evaluation will be conducted to examine: to what extent it is possible to implement problem-solving therapy according to the protocol; the relationship between the key elements of problem-solving intervention and the effect outcome; how the participants perceive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* employed women and men aged 18-59, short-term sick leave (i.e. a minimum of 2 weeks and a maximum of 12 weeks) due to mild to moderate depression, anxiety or adjustment disorder (F 32, F 41, F 43) as the primary reason for sick leave, diagnosed by a general practitioner (GP) or physician according to the Swedish version of international statistical classification of diseases and related health problems - tenth revision (ICD-10) contact with a GP or physician at a primary health care center in the vestra gotaland region.

Exclusion Criteria:

* Severe depression, other severe mental disorders, i.e. psychotic or bipolar disorders; pregnancy, somatic complaints or disorders that will influence work ability; not able to read, write and understand Swedish.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Change in total registered sickness absenteeism in number of days from baseline during the 18 month follow-up. | At baseline and 18 months after baseline.
  Change in total registered sickness absenteeism in number of days from baseline during the 18 months follow-up (including sickness benefit, sickness and activity compensation, disability pension). Data from the Social Insurance Agency's register MiDAS.
  The analyses will be repeated for outcomes on registered sickness absence at a three-year follow-up.

SECONDARY OUTCOMES:
Change from baseline in registered part-time sickness absenteeism during the 18 months follow-up | From baseline to 18 months after baseline.
  Change from baseline in registered partial sickness absenteeism (25/50/75% of full-time sickness absenteeism) during a follow-up period of 18 months. Change in registered sickness absenteeism will be calculated from baseline until the 18 months follow-up in number of days on part-time sick leave (25/50/75% of full-time sick leave). Data from the Social Insurance Agency's register MiDAS.
Change from baseline in return to work during a period of 18 months. | From baseline to 18 months after baseline.
  Change from baseline in return to work during a follow-up of 18 months. Return to work will be calculated from baseline data until the individual returns to work in ordinary hours during an uninterrupted period of at least four weeks.
Episodes of sickness absenteeism after full-time return to work | From baseline during 18 months follow-up.
  Episodes of sick leave after full-time return to work (i.e. work in ordinary hours during an uninterrupted period of at least four weeks) will be calculated from baseline until the 18 months follow-up by registered sickness absenteeism.
Change in total registered sick leave from baseline to 36 month follow-up. | Change in total registered sick leave from baseline to 36 month follow-up.
  Change in total registered sickness absenteeism at baseline and during the 36 months follow-up (including sickness benefit, sickness and activity compensation, disability pension). Data from the Social Insurance Agency's register MiDAS.
Possible interaction effects | Change from baseline and 6, 12 and 18 months after study inclusion.
  Possible interaction effects on the primary and secondary outcomes for (1) gender x treatment, and (2) number of sessions with rehabilitation coordinator x treatment will be checked for and if statistically significant subgroup analyses will be considered.
Self-reported short-term sickness absenteeism | From baseline to 12 months after baseline.
  Change in self-reported sickness absenteeism from baseline during the 12 month follow-up. Self-reported data collected every fourth week during the 12 months. These self-reported data cover shorter spells of sickness absenteeism (i.e. ≤14 consecutive days) that is not covered by the Social Insurance Agency's register.
Change from baseline in self-reported part-time sickness absenteeism during the 12 months follow-up | From baseline to 12 months after baseline.
  Change from baseline in self-reported partial sickness absenteeism (25/50/75% of full-time sickness absenteeism) during a follow-up period of 12 months. Change in self-reported sickness absenteeism will be calculated from baseline until the 12 months follow-up in number of days on part-time sick leave (25/50/75% of full-time sick leave).
Change from baseline in return to work during a period of 12 months. | From baseline to 12 months after baseline.
  Change from baseline in self-reported return to work during a follow-up of 12 months. Return to work will be calculated from baseline data until the individual returns to work in ordinary hours during an uninterrupted period of at least four weeks. Self-reported data obtained every fourth week during a period of 12 months.
Episodes of self-reported sickness absenteeism after full-time return to work. | From baseline during 12 months follow-up.
  Episodes of self-reported sickness absenteeism after full-time return to work (i.e. work in ordinary hours during an uninterrupted period of at least four weeks) will be calculated from baseline until the 12 months follow-up by self-reported sickness absenteeism.
Reduction of symptoms related to common mental disorders Hospital Anxiety and Depression scale | Baseline and 6 and 12 months after study inclusion.
  Hospital Anxiety and Depression Scale will be used to assess symptoms of anxiety (seven items) and depression (seven items). Each item is scored on a 4-point Likert scale indicating the extent to which an item was experienced in the past week. Response format from 0 to 3.
Reduction of symptoms related to common mental disorders Self-reported exhaustion | Baseline and 6 and 12 months after study inclusion.
  Institute of Stress Medicine's instrument for self-reported exhaustion: Change from baseline in self-reported exhaustion as measured by the Institute of Stress Medicine's instrument. Three items with the response format yes/no and one item with response format from 0 to 2.
Reduction of symptoms related to common mental disorders Karolinska Sleep Questionnaire | Baseline and 6 and 12 months after study inclusion.
  Karolinska Sleep Questionnaire, Insomnia subscale will be used for assessing insomnia problems. The subscale includes four items. Each item is scored on a 6 point scale ranging from 0 (never) to 5 (always) indicating to what extent an item was experienced in the last three months. Change from baseline in self-reported sleep problems.
Sickness presenteeism | Baseline and after 6 and 12 months after study inclusion.
  Sickness presenteeism will be measured with a single question, response format 1-4.
Work ability index (WAI) | Baseline and 6 and 12 months after study inclusion.
  WAI: change from baseline and after 6 and 12 months after study inclusion, self-reported work ability is assessed by 2 items from WAI (with the response format 1 - 5). These questions measures the perceived work capacity in relation to the physical (1 item) and the mental (1 item) demands of the work.
Work performance impairment due to health problems | Will be assessed at baseline and once a month during a 12-month follow-up period.
  Work performance due to health problems will be measured by a question from one of the items included in the Work Productivity Impairment - General Health Questionnaire (the response format is 0-10).
Work performance impairment due to problems in the working environment | Will be assessed at baseline and once a month during a 12-month follow-up period.
  Work performance due to problems in the working environment will be measured by a question from one of the items included in the Work Productivity Impairment - General Health Questionnaire (the response format is 0-10).
Demand-control-support | Baseline and after 6 and 12 months after study inclusion.
  Demand-control-support model: Change from baseline and after 6 and 12 months after study inclusion, response format from 1 to 4. Prognostic variable.
Return-to-work self-efficacy | Change from baseline and 6 and 12 months after study inclusion.
  Return-to-work self-efficacy will be measured by a question with the response format from 0 to 10. Prognostic variable.
Ongoing conflict with the superior | Change from baseline at 6 and 12 months after study inclusion.
  Ongoing conflict with the superior is measured by one item. The item is scored on a 3 point Likert-type scale ranging from 0 (never) to 3 (often or always). Prognostic variable.
Perceived loss of control over work tasks | Change from baseline at 6 and 12 months after study inclusion.
  Perceived loss of control over work tasks is measured by one item. The item is scored on a Likert-type scales with 5 response options ranging from 0 (never or almost never) to 4 (very often or always). Prognostic variable.
Conflict between employee's values and how the work actually is done | Change from baseline at 6 and 12 months after study inclusion.
  Conflict between employee's values and how the work actually is done is measured by three items. Each item is scored on a Likert-type scale5 response options ranging from 0 (never or almost never) to 4 (very often or always). Prognostic variable.
Job strain | Change from baseline at 6 and 12 months after study inclusion.
  Job strain (emotional and psychological demands) will be assessed by four items from Copenhagen psychosocial questionnaire, response format is likert-type scales with 5 response options. Prognostic variable.
Participants' satisfaction | Will be assessed at 6 months after intervention.
  Participants' satisfaction and experiences with their participation in the intervention or care as usual will be assessed at 6 months after completed intervention, as a part of the process evaluation. Self-reported questionnaire with ten items, response format from 0 to 10 or yes/no/do not know.
The rehabilitation coordinators' adherence to the intervention. | Assessed immediately upon completion of intervention.
  The rehabilitation coordinators' adherence to the intervention is measured by a single item with the response format from 1 to 5.
Health related quality of life | Will be measured at baseline, 6 and 12 months follow-up
  Health related quality of life will be measured with European Quality of Life 5 Dimensions questionnaire (EQ5D). The response format is a 3-level scale, with higher levels indicating severity.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Björk Brämberg, PhD, Principal Investigator — Karolinska Institute, Unit of intervention and implementation research
Locations (2):
- Sweden (2):
  - Primary health care, Gothenburg, Region Västra Götaland
  - Elisabeth Björk Brämberg, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data available. In line with the study's ethical approval, data may only be made available after reasonable request to the principal investigator, and after decision by the Swedish Ethical Review Authority.
Supporting Information: Study Protocol
Access Criteria: There is a plan to make IPD and related data available. In line with the study's ethical approval, data may only be made available after reasonable request to the principal investigator, and after decision by the Swedish Ethical Review Authority.

REFERENCES:
- [Derived] Eklund A, Karlsson I, Bergstrom G, Lisa H, Elisabeth BB. The effectiveness of a problem-solving intervention with workplace involvement on self-reported sick leave, psychological symptoms and work ability: a cluster randomised clinical trial. BMC Public Health. 2024 Nov 5;24(1):3052. doi: 10.1186/s12889-024-20564-z. PMID 39501245
- [Derived] Karlsson I, Frantz A, Axen I, Bergstrom G, Bultmann U, Finnes A, Holmgren K, Kwak L, Bjork Bramberg E. Is a Problem-Solving Intervention with Workplace Involvement for Employees on Sickness Absence Due to Common Mental Disorders More Effective, than Care as Usual, in Reducing Sickness Absence Days? Results of a Cluster-Randomised Controlled Trial in Primary Health Care. J Occup Rehabil. 2025 Sep;35(3):615-624. doi: 10.1007/s10926-024-10229-4. Epub 2024 Aug 7. PMID 39110387
- [Derived] Toropova A, Bjork Bramberg E, Bergstrom G. Return to Work Trajectories of Swedish Employees on Sick-Leave Due to Common Mental Disorders. J Occup Rehabil. 2025 Sep;35(3):479-490. doi: 10.1007/s10926-024-10216-9. Epub 2024 Jun 22. PMID 38907784
- [Derived] Holmlund L, Ljungberg HT, Bultmann U, Bramberg EB. Navigating work and life- a qualitative exploration of managers' and employees' views of return-to-work after sick leave due to common mental disorders. BMC Public Health. 2024 Feb 5;24(1):372. doi: 10.1186/s12889-024-17765-x. PMID 38317150
- [Derived] Bjork Bramberg E, Holmgren K, Bultmann U, Gyllensten H, Hagberg J, Sandman L, Bergstrom G. Increasing return-to-work among people on sick leave due to common mental disorders: design of a cluster-randomized controlled trial of a problem-solving intervention versus care-as-usual conducted in the Swedish primary health care system (PROSA). BMC Public Health. 2018 Jul 18;18(1):889. doi: 10.1186/s12889-018-5816-8. PMID 30021545